CLINICAL TRIAL: NCT02563093
Title: Safety and Immunogenicity Among Adults of Fluzone® Quadrivalent, Fluzone® Intradermal Quadrivalent, and Fluzone® High-Dose, Influenza Vaccines, 2015-2016 Formulations
Brief Title: Study of Fluzone® Quadrivalent, Fluzone® Intradermal Quadrivalent, and Fluzone® High-Dose, Influenza Vaccines in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC57; U1111-1161-2491 (Other: WHO)
Record Dates: First submitted 2015-09-28; First posted 2015-09-29 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-10

CONDITIONS: Influenza
Keywords: Influenza; Fluzone® Quadrivalent, Influenza Vaccine; Fluzone® Intradermal Quadrivalent, Influenza Vaccine; Fluzone® High Dose, Influenza Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Study Group 1 (Experimental): Adults 18 to < 65 years of age randomly assigned to receive an intramuscular injection of one dose of Fluzone Quadrivalent vaccine
  Interventions: Biological: Fluzone Quadrivalent vaccine, 2015-2016 formulation, No Preservative
- Study Group 2 (Experimental): Adults 18 to < 65 years of age randomly assigned to receive an intradermal injection of one dose of Fluzone Intradermal Quadrivalent vaccine
  Interventions: Biological: Fluzone Intradermal Quadrivalent vaccine, 2015-2016 formulation
- Study Group 3 (Experimental): Adults ≥ 65 years of age randomly assigned to receive an intramuscular injection of one dose of Fluzone Quadrivalent vaccine
  Interventions: Biological: Fluzone Quadrivalent vaccine, 2015-2016 formulation, No Preservative
- Study Group 4 (Experimental): Adults ≥ 65 years of age randomly assigned to receive an intramuscular injection of one dose of Fluzone High-Dose vaccine
  Interventions: Biological: Fluzone High-Dose vaccine, 2015-2016 formulation

INTERVENTIONS:
Biological: Fluzone Quadrivalent vaccine, 2015-2016 formulation, No Preservative — 0.5 mL, Intramuscular (IM)
  Other Names: Fluzone® Quadrivalent, Influenza Vaccine
  Arms: Study Group 1
Biological: Fluzone Intradermal Quadrivalent vaccine, 2015-2016 formulation — 0.1 mL, Intradermal
  Other Names: Fluzone® Intradermal Quadrivalent, Influenza Vaccine
  Arms: Study Group 2
Biological: Fluzone Quadrivalent vaccine, 2015-2016 formulation, No Preservative — 0.5 mL, Intramuscular
  Other Names: Fluzone® Quadrivalent, Influenza Vaccine
  Arms: Study Group 3
Biological: Fluzone High-Dose vaccine, 2015-2016 formulation — 0.5 mL, Intramuscular
  Other Names: Fluzone® High-Dose, Influenza Vaccine
  Arms: Study Group 4

SUMMARY:
The aim of the study is to evaluate the safety and immunogenicity of the 2015-2016 formulations of Fluzone Quadrivalent and Fluzone Intradermal Quadrivalent vaccines in adults 18 to < 65 years of age, and of the 2015-2016 formulations of Fluzone Quadrivalent and Fluzone High-Dose vaccines in adults ≥ 65 years of age.

Primary Objective:

- To describe the safety of the 2015-2016 formulations of Fluzone Quadrivalent and Fluzone Intradermal Quadrivalent vaccines in adults 18 to < 65 years of age and the safety of the 2015-2016 formulations of Fluzone Quadrivalent and Fluzone High-Dose vaccines in adults ≥ 65 years of age.

Observational Objectives:

* To describe the immunogenicity of the 2015-2016 formulations of Fluzone Quadrivalent and Fluzone Intradermal Quadrivalent vaccines in adults 18 to < 65 years of age and the immunogenicity of the 2015-2016 formulations of Fluzone Quadrivalent and Fluzone High-Dose vaccines in adults ≥ 65 years of age.
* To evaluate the compliance, in terms of immunogenicity, of each study vaccine (Fluzone Quadrivalent, Fluzone Intradermal Quadrivalent, and Fluzone High-Dose) in the applicable age group with the historical requirements of the Committee for Human Medicinal Products (CHMP) Note for Guidance (NfG) Committee for Propriety Medicinal Products (CPMP) - CHMP NfG CPMP/BWP/214/96.

DETAILED DESCRIPTION:
Adults age 18 to < 65 years will be randomly assigned to receive either Fluzone Quadrivalent or Fluzone Intradermal Quadrivalent vaccine and adults age ≥ 65 years will be randomly assigned to receive either Fluzone Quadrivalent or Fluzone High-Dose vaccine. All subjects will receive a single dose of their randomly assigned vaccine.

They will be followed from Visit 1 to Visit 2 for evaluation of safety outcomes. Solicited adverse reactions will be collected for 7 days after vaccination. Unsolicited non-serious adverse events (AEs) and serious adverse events (SAEs) will be collected from Visit 1 to Visit 2.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age on the day of inclusion
* Informed consent form has been signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* History of serious adverse reaction to any influenza vaccine
* Receipt of any vaccine within 30 days before receiving study vaccine, or plans to receive another vaccine before Visit 2
* Participation in another interventional clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 30 days preceding the first study vaccination or during the course of the study, unless no intervention for the other study occurred within the 30 days prior to the first study vaccination and none are planned before the subject would complete safety surveillance for the present study
* Thrombocytopenia, which may be a contraindication for intramuscular vaccination, at the discretion of the Investigator
* Prior vaccination with any 2015-2016 formulation of influenza vaccine
* Known systemic hypersensitivity to eggs, chicken proteins, or any of the vaccine components, or a history of a life-threatening reaction to Fluzone Quadrivalent, Fluzone Intradermal Quadrivalent, or Fluzone High-Dose vaccine or to a vaccine containing any of the same substances (the complete list of vaccine components is included in the Prescribing Information)
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, which may be a contraindication for intramuscular vaccination, at the discretion of the Investigator
* Subject is pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination and until at least 4 weeks after vaccination)
* Any condition that in the opinion of the Investigator would pose a health risk to the subject if enrolled or could interfere with the evaluation of the vaccine
* Personal history of Guillain-Barré syndrome
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion
* Seropositivity for human immunodeficiency virus, hepatitis B, or hepatitis C, as reported by the subject.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol or drug addiction that, in the opinion of the Investigator, might interfere with the ability to comply with trial procedures
* Moderate or severe acute illness/infection (according to Investigator judgment) or febrile illness (temperature ≥ 100.4°F) on the day of vaccination. A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as an Investigator or employee of an Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of an Investigator or employee with direct involvement in the proposed study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (4):
- United States (4):
  - Santa Rosa, California
  - Council Bluffs, Iowa
  - Metairie, Louisiana
  - Cincinnati, Ohio

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 28 September 2015 to 03 November 2015 at 4 clinic centers in the United States.
Pre-assignment Details: A total of 208 participants who met all of the inclusion criteria and no exclusion criteria were enrolled and vaccinated.
Groups:
- Fluzone Quadrivalent Vaccine (18 to < 65 Years): Adults 18 to < 65 years of age who received an intramuscular injection of a dose of Fluzone Quadrivalent vaccine
- Fluzone Quadrivalent Intradermal Vaccine (18 to < 65 Years): Adults 18 to < 65 years of age who received an intradermal injection of a dose of Fluzone Intradermal Quadrivalent vaccine
- Fluzone Quadrivalent Vaccine (≥ 65 Years): Adults ≥ 65 years of age who received an intramuscular injection of a dose of Fluzone Quadrivalent vaccine
- Fluzone High-Dose Vaccine (≥ 65 Years): Adults ≥ 65 years of age who received an intramuscular injection of a dose of Fluzone High-Dose vaccine
Period: Overall Study
Arm/Group | Fluzone Quadrivalent Vaccine (18 to < 65 Years) | Fluzone Quadrivalent Intradermal Vaccine (18 to < 65 Years) | Fluzone Quadrivalent Vaccine (≥ 65 Years) | Fluzone High-Dose Vaccine (≥ 65 Years)
Started | 52 | 52 | 53 | 51
Completed | 52 | 52 | 53 | 51
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fluzone Quadrivalent Intradermal Vaccine: Adults 18 to < 65 years of age who received an intradermal injection of a dose of Fluzone Intradermal Quadrivalent vaccine
- Fluzone High-Dose Vaccine: Adults ≥ 65 years of age who received an intramuscular injection of a dose of Fluzone High-Dose vaccine
- Total: Total of all reporting groups
Arm/Group | Fluzone Quadrivalent Vaccine (18 to < 65 Years) | Fluzone Quadrivalent Intradermal Vaccine | Fluzone Quadrivalent Vaccine (≥ 65 Years) | Fluzone High-Dose Vaccine | Total
Number analyzed (Participants) | 52 | 52 | 53 | 51 | 208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 52 | 52 | 0 | 0 | 104
  >=65 years | 0 | 0 | 53 | 51 | 104
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.4 (13.5) | 43.4 (14.7) | 72.8 (5.2) | 74.2 (6.2) | 59.2 (17.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 39 | 28 | 26 | 130
  Male | 15 | 13 | 25 | 25 | 78
Region of Enrollment [Number; unit: Participants]
  United States | 52 | 52 | 53 | 51 | 208

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Injection-Site or Systemic Reactions After Receipt of the 2015-2016 Formulation of Fluzone Quadrivalent, Fluzone Intradermal Quadrivalent, or Fluzone High-Dose Vaccine
Description: Solicited injection-site reactions: Pain, Erythema, Swelling, Induration, and Ecchymosis. Solicited systemic reactions: Fever, Headache, Malaise, Myalgia, and Shivering. Grade 3 solicited injection-site reactions: Pain, Significant; prevents daily activity. Erythema, Swelling, Induration, and Ecchymosis >100 mm. Grade 3 solicited systemic reactions: Fever, ≥ 39.0°C or ≥ 102.1°F; Headache, Malaise, Myalgia, and Shivering, Significant; prevents daily activity.
  A participant (18 to < 65 Years) who was randomly assigned to receive Fluzone Intradermal Quadrivalent vaccine received Fluzone Quadrivalent vaccine instead; this participant was excluded from the Per-protocol analysis Set and was included in the Fluzone Quadrivalent vaccine Group in the Safety Analysis Set and the assigned group in the Full Analysis Set.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: The vaccine safety outcomes were assessed in the Safety Analysis Set. A participant (18 to < 65 Years) who was assigned to receive Fluzone Intradermal Quadrivalent vaccine received Fluzone Quadrivalent vaccine instead; this participant was included in the Fluzone Quadrivalent vaccine (18 to < 65 Years) group in the Safety Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Fluzone Quadrivalent Vaccine (18 to < 65 Years) | Fluzone Quadrivalent Intradermal Vaccine (18 to < 65 Years) | Fluzone Quadrivalent Vaccine (≥ 65 Years) | Fluzone High-Dose Vaccine (≥ 65 Years)
Number analyzed (Participants) | 53 | 51 | 53 | 51
Participants
  Injection-site Pain (N=53, 51, 53, 51) | 29 | 29 | 15 | 22
  Grade 3 Injection-site Pain (N=53, 51, 53, 51) | 0 | 0 | 1 | 0
  Injection-site Erythema (N=53, 51, 53, 51) | 1 | 17 | 0 | 7
  Grade 3 Injection-site Erythema (N=53, 51, 53, 51) | 0 | 0 | 0 | 0
  Injection-site Swelling (N=53, 51, 53, 51) | 1 | 10 | 0 | 3
  Grade 3 Injection-site Swelling (N=53, 51, 53, 51) | 0 | 0 | 0 | 0
  Injection-site Induration (N=53, 51, 53, 51) | 1 | 6 | 0 | 1
  Grade 3 Injection-site Induration (N=53,51,53,51) | 0 | 0 | 0 | 0
  Injection-site Ecchymosis (N=53, 51, 53, 51) | 1 | 1 | 0 | 2
  Grade 3 Injection-site Ecchymosis (N=53,51,53,51) | 0 | 0 | 0 | 0
  Fever (N=52, 51, 53, 51) | 0 | 0 | 0 | 0
  Grade 3 Fever (N=52, 51, 53, 51) | 0 | 0 | 0 | 0
  Headache (N=53, 51, 53, 51) | 13 | 12 | 9 | 6
  Grade 3 Headache (N=53, 51, 53, 51) | 0 | 2 | 1 | 0
  Malaise (N=53, 51, 53, 51) | 7 | 11 | 10 | 6
  Grade 3 Malaise (N=53, 51, 53, 51) | 0 | 2 | 0 | 0
  Myalgia (N=53, 51, 53, 51) | 15 | 11 | 9 | 13
  Grade 3 Myalgia (N=53, 51, 53, 51) | 1 | 1 | 0 | 0
  Shivering (N=53, 51, 53, 51) | 6 | 0 | 1 | 0
  Grade 3 Shivering (N=53, 51, 53, 51) | 0 | 0 | 0 | 0

2. Secondary Outcome: Geometric Mean Titers of Influenza Antibodies Pre- and Post-Vaccination With the 2015-2016 Formulation of Fluzone Quadrivalent, Fluzone Intradermal Quadrivalent, or Fluzone High-Dose Vaccine
Description: Anti-influenza antibodies were measured using an hemagglutination inhibition assay.
Time Frame: Day 0 (pre-vaccination) and 21 days post-vaccination
Population: Anti-influenza antibodies were assessed in the Per-protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilutions)
Arm/Group | Fluzone Quadrivalent Vaccine (18 to < 65 Years) | Fluzone Quadrivalent Intradermal Vaccine (18 to < 65 Years) | Fluzone Quadrivalent Vaccine (≥ 65 Years) | Fluzone High-Dose Vaccine (≥ 65 Years)
Number analyzed (Participants) | 51 | 50 | 53 | 51
Titers (1/dilutions)
  A/H1N1; Pre-vaccination (N=51,50,53,51) | 274 [173 to 433] | 196 [134 to 286] | 160 [109 to 234] | 62.2 [44.4 to 87.3]
  A/H1N1; Post-vaccination (N=51,50,53,51) | 764 [564 to 1034] | 631 [435 to 915] | 283 [196 to 407] | 324 [242 to 435]
  A/H3N2; Pre-vaccination (N=51,50,53,51) | 49.4 [32.0 to 76.2] | 61.9 [44.4 to 86.3] | 48.0 [34.4 to 67.0] | 50.1 [36.4 to 68.7]
  A/H3N2; Post-vaccination (N=51,50,53,51) | 1051 [687 to 1609] | 1033 [717 to 1488] | 379 [248 to 580] | 769 [517 to 1143]
  B Yamagata; Pre-vaccination (N=51,50,53,51) | 186 [118 to 293] | 307 [208 to 454] | 208 [147 to 293] | 134 [101 to 179]
  B Yamagata; Post-vaccination (N=51,50,53,51) | 881 [581 to 1336] | 1099 [822 to 1469] | 438 [311 to 617] | 471 [352 to 632]
  B Victoria; Pre-vaccination (N=51,50,53,0) | 234 [161 to 340] | 290 [213 to 397] | 178 [122 to 258] | NA [NA to NA] — B Victoria Influenza antigen not in administered vaccine for this group
  B Victoria; Post-vaccination (N=51,50,53,0) | 1237 [901 to 1700] | 844 [621 to 1149] | 355 [260 to 485] | NA [NA to NA] — B Victoria Influenza antigen not in administered vaccine for this group

3. Secondary Outcome: Number of Participants Achieving Seroprotection Pre and Post-Vaccination With the 2015-2016 Formulation of Fluzone Quadrivalent, Fluzone Intradermal Quadrivalent, or Fluzone High-Dose Vaccine
Description: Anti-influenza antibodies were measured using an hemagglutination inhibition assay. Seroprotection was defined as the number of participants with a titer ≥ 40 (1/dilution) at pre-vaccination and 21 days post-vaccination.
Time Frame: Day 0 (Pre-vaccination) and 21 days post-vaccination
Population: Anti-influenza antibodies were assessed in the Per-protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Fluzone Quadrivalent Vaccine (18 to < 65 Years) | Fluzone Quadrivalent Intradermal Vaccine (18 to < 65 Years) | Fluzone Quadrivalent Vaccine (≥ 65 Years) | Fluzone High-Dose Vaccine (≥ 65 Years)
Number analyzed (Participants) | 51 | 50 | 53 | 51
Participants
  A/H1N1; Pre-vaccination (N=51,50,53,51) | 45 | 47 | 47 | 38
  A/H1N1; Post-vaccination (N=51,50,53,51) | 51 | 50 | 50 | 50
  A/H3N2; Pre-vaccination (N=51,50,53,51) | 32 | 35 | 36 | 28
  A/H3N2; Post vaccination (N=51,50,53,51) | 50 | 50 | 50 | 51
  B Yamagata; Pre-vaccination (N=51,50,53,51) | 41 | 48 | 51 | 48
  B Yamagata; Post-vaccination (N=51,50,53,51) | 51 | 50 | 53 | 51
  B Victoria; Pre-vaccination (N=51,50,53,0) | 47 | 49 | 49 | NA — B Victoria Influenza antigen not in administered vaccine for this group
  B Victoria; Post-vaccination (N=51,50,53,0) | 51 | 49 | 53 | NA — B Victoria Influenza antigen not in administered vaccine for this group

4. Secondary Outcome: Number of Participants Achieving Seroconversion Following Vaccination With the 2015-2016 Formulation of Fluzone Quadrivalent, Fluzone Intradermal Quadrivalent, or Fluzone High-Dose Vaccine
Description: Anti-influenza antibodies were measured using an hemagglutination inhibition assay. Seroconversion was defined as either a pre-vaccination titer < 1:10 and a post-vaccination titer ≥ 1:40, or a pre-vaccination titer ≥ 1:10 and a ≥ 4-fold increase in titer post-vaccination.
Time Frame: 21 days post-vaccination
Population: Anti-influenza antibodies were assessed in the Per-protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Fluzone Quadrivalent Vaccine (18 to < 65 Years) | Fluzone Quadrivalent Intradermal Vaccine (18 to < 65 Years) | Fluzone Quadrivalent Vaccine (≥ 65 Years) | Fluzone High-Dose Vaccine (≥ 65 Years)
Number analyzed (Participants) | 51 | 50 | 53 | 51
Participants
  A/H1N1 (N=51,50,53,51) | 15 | 17 | 9 | 27
  A/H3N2 (N=51,50,53,51) | 44 | 42 | 35 | 44
  B Yamagata (N=51,50,53,51) | 29 | 24 | 13 | 23
  B Victoria (N=51,50,53,0) | 27 | 15 | 9 | NA — B Victoria Influenza antigen not in administered vaccine for this group

5. Secondary Outcome: Geometric Mean Titer Ratios of Influenza Antibodies Post-Vaccination With the 2015-2016 Formulation of Fluzone Quadrivalent, Fluzone Intradermal Quadrivalent, or Fluzone High-Dose Vaccine
Description: Anti-influenza antibodies were measured using an hemagglutination inhibition assay.
Time Frame: 21 days post-vaccination
Population: Anti-influenza antibodies were assessed in the Per-protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratio
Arm/Group | Fluzone Quadrivalent Vaccine (18 to < 65 Years) | Fluzone Quadrivalent Intradermal Vaccine (18 to < 65 Years) | Fluzone Quadrivalent Vaccine (≥ 65 Years) | Fluzone High-Dose Vaccine (≥ 65 Years)
Number analyzed (Participants) | 51 | 50 | 53 | 51
Titer ratio
  A/H1N1 (N=51,50,53,51) | 2.72 [1.92 to 3.84] | 3.18 [2.25 to 4.49] | 1.77 [1.38 to 2.26] | 5.07 [3.50 to 7.35]
  A/H3N2 (N=51,50,53,51) | 19.4 [12.5 to 29.9] | 16.4 [10.4 to 26.1] | 7.49 [4.97 to 11.3] | 15.2 [10.2 to 22.5]
  B Yamagata (N=51,50,53,51) | 4.74 [3.22 to 6.98] | 3.58 [2.52 to 5.09] | 2.11 [1.60 to 2.78] | 3.52 [2.59 to 4.76]
  B Victoria (N=51,50,53,0) | 5.29 [3.54 to 7.89] | 2.87 [2.15 to 3.83] | 1.97 [1.52 to 2.57] | NA [NA to NA] — B Victoria Influenza antigen not in administered vaccine for this group

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 up to Day 21 post-vaccination.
Description: A participant (18 to < 65 Years) who was randomly assigned to receive Fluzone Intradermal Quadrivalent vaccine received Fluzone Quadrivalent vaccine instead; this participant was included in the Fluzone Quadrivalent vaccine (18 to < 65 Years) Group in the Safety Analysis Set.
Arm/Group | Fluzone Quadrivalent Vaccine (18 to < 65 Years) | Fluzone Quadrivalent Intradermal Vaccine (18 to < 65 Years) | Fluzone Quadrivalent Vaccine (≥ 65 Years) | Fluzone High-Dose Vaccine (≥ 65 Years)
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/51 | 0/53 | 1/51
Other Adverse Events (participants affected / at risk) | 29/53 | 29/51 | 15/53 | 22/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone Quadrivalent Vaccine (18 to < 65 Years) (N=53) | Fluzone Quadrivalent Intradermal Vaccine (18 to < 65 Years) (N=51) | Fluzone Quadrivalent Vaccine (≥ 65 Years) (N=53) | Fluzone High-Dose Vaccine (≥ 65 Years) (N=51)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone Quadrivalent Vaccine (18 to < 65 Years) (N=53) | Fluzone Quadrivalent Intradermal Vaccine (18 to < 65 Years) (N=51) | Fluzone Quadrivalent Vaccine (≥ 65 Years) (N=53) | Fluzone High-Dose Vaccine (≥ 65 Years) (N=51)
Injection site Pruritus (General disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Injection site Pain (General disorders) | 29 (29) | 29 (29) | 15 (15) | 22 (22)
Injection site Erythema (General disorders) | 1 (1) | 17 (17) | 0 (0) | 7 (7)
Injection site Swelling (General disorders) | 1 (1) | 10 (10) | 0 (0) | 3 (3)
Injection site Induration (General disorders) | 1 (1) | 6 (6) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 13 (13) | 12 (12) | 9 (9) | 6 (6)
Malaise (General disorders) | 7 (7) | 11 (11) | 10 (10) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (15) | 11 (11) | 9 (9) | 13 (13)
Shivering (General disorders) | 6 (6) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications